CLINICAL TRIAL: NCT05307406
Title: A First-in-Human Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Exploratory Markers of Efficacy for XAB05 in Healthy Subjects
Brief Title: A First-in-Human Study With XAB05 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xenothera SAS (Industry)
Collaborators: QPS Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XT-2102
Record Dates: First submitted 2022-02-17; First posted 2022-04-01 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XAB05 (Experimental): Single ascending dose from 0.25 mg/kg up to 20mg/kg IV infusion
  Interventions: Biological: Experimental
- Placebo (Placebo Comparator): Single IV infusion
  Interventions: Biological: Experimental

INTERVENTIONS:
Biological: Experimental — Participants will receive a single IV infusion in a double blind manner

SUMMARY:
This study is a randomized, placebo-controlled, first in human, single ascending dose Phase 1 study

DETAILED DESCRIPTION:
This study is a First in Human (FIH) single ascending dose study with XAB05 to evaluate safety, tolerability, PK and exploratory markers of efficacy for XAB05 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* .The subject must understand the nature of the study and must provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-related procedures.

  2. Healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG recording. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied, may be included only if, in the opinion of the Investigator, the finding is (a) unlikely to introduce additional risk to the subject, (b) will not interfere with study procedures or confound study results, and (c) is not otherwise exclusionary (see Exclusion Criteria).

  3. The subject is a male or female, aged 18 to 65 years, inclusive, at Screening.

  4. The subject weighs at least 50 kg and has a BMI between 18.0 and 34.0 kg/m2, inclusive, at Screening and on Day -1.

  5. Women of child-bearing potential must agree not to attempt to become pregnant and to use a highly effective form of hormonal (oral contraception, a hormonal implant, hormonal injection or hormonal intra-uterine devices) or non-hormonal (non-hormonal intra-uterine device/system in combination with a barrier method (e.g. condom, diaphragm, cervical cap with spermicide)) birth control or abstinence during the study and for 90 days after the (last) study drug administration. Postmenopausal women must have had ≥12 months of spontaneous amenorrhea (with documented follicle-stimulating hormone (FSH) ≥30 mIU/mL). Surgically sterile women are defined as those who have had a hysterectomy, bilateral ovariectomy, or bilateral tubal ligation. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound. All women must have a negative pregnancy test result at Screening and on Day -1.

Exclusion Criteria:

* 1. The subject has history or evidence of clinically significant hematologic, dermatologic, neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic including difficulty voiding, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the subject to participate or potentially confound the study results, or which, in the investigator's opinion, makes subjects unsuitable for the study.

  2. The subject has a significant history of allergies, as determined by the Principal Investigator.

  3. The subject is taking antihistamines, NSAIDs, or mast cell stabilizers (e.g. disodium cromoglycate) and is unable to stop taking these medications from 7 days prior to Day 1.

  4. The subject has received any prescription or non-prescription drugs (including steroids and COVID-19 vaccination, but excluding paracetamol, oral contraception, a hormonal implant or hormonal intra-uterine devices), vitamins and herbal remedies (including St John's Wort), within 14 days or 5 half-lives (whichever is longer) prior to Day -1.

  5. A clinically significant abnormality on physical examination, ECG, or laboratory evaluations at Screening or between Screening and study drug administration.

  6. The subject has a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 45 to 90 mm Hg for diastolic, confirmed on repeat testing at Screening and on Day -1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters: physical examination | From screening through study completion, up to 30 days
  Number of clinically relevant findings during inspection, percussion, palpation, and auscultation.
Safety and tolerability parameters: Adverse events (AEs) | From screening through study completion, up to 30 days
  Number of adverse events (AEs)
Safety and tolerability parameters :infusion site reactions/local tolerability | From screening through study completion, up to 30 days
  Incidence of infusion site reactions/local tolerability
Safety and tolerability parameters: clinical laboratory values | From screening through study completion, up to 30 days
  Number of clinically significant laboratory abnormalities
Safety and tolerability parameters:vital signs - Blood pressure value | From screening through study completion, up to 30 days
  Blood pressure (mm Hg)
Safety and tolerability parameters:vital signs - Pulse value | From screening through study completion, up to 30 days
  pulse rate
Safety and tolerability parameters:vital signs -repiratory value | From screening through study completion, up to 30 days
  respiration rate
Safety and tolerability parameters:vital signs -temperature | From screening through study completion, up to 30 days
  temporal body temperature
Safety and tolerability parameters: electrocardiogram (ECG): | From screening through study completion, up to 30 days
  Number of Clinically significant abnormal findings recorded by investigator based on HR, PR, QRS, and QT values of ECG

SECONDARY OUTCOMES:
PK parameters for XAB05 : Cmax | From treatment day through study completion, up to 30 days
  Maximal Observed concentration (Cmax)
PK parameters for XAB05: tmax | From treatment day through study completion, up to 30 days
  Time to Cmax
PK parameters for XAB05 :Ceoi | From treatment day through study completion, up to 30 days
  Concentration at the end of infusion
PK parameters for XAB05 : t1/2 | From treatment day through study completion, up to 30 days
  Terminal elimination half-life of the drug
PK parameters for XAB05 : AUC0-t | From treatment day through study completion, up to 30 days
  Area under the concentration-time curve up to the last measurable concentration
PK parameters for XAB05 :AUC0-inf | From treatment day through study completion, up to 30 days
  Area under the concentration-time curve to infinite time
PK parameters for XAB05: CL | From treatment day through study completion, up to 30 days
  Clearance of the drug
PK parameters for XAB05 : Vz | From treatment day through study completion, up to 30 days
  Volume of distribution
Immunogenicity parameters | From treatment day through study completion, up to 30 days
  concentration of anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Khadid Abd-Elaziz, MD, Principal Investigator — QPS Netherlands B.V.
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands